CLINICAL TRIAL: NCT07067372
Title: Clinical Study on the Safety and Efficacy of FireMagic™ Magbot Ablation Catheter for Rapid Arrhythmia
Brief Title: Clinical Study on the Safety and Efficacy of a New Magnetic Navigation Radiofrequency Ablation Catheter for Rapid Arrhythmia
Acronym: Rapid arrhythm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gao Henggan, Shanghai MicroPort EP MedTech Co., Ltd., Ruijin-Hainan Hospital Shanghai Jiao Tong University School Of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240710
Record Dates: First submitted 2025-06-20; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Rapid Arrhythmia; PFA; Symptomatic Supraventricular Tachycardia
Keywords: Paroxysmal atrial fibrillation; Symptomatic supraventricular tachycardia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical study on the safety and efficacy ofFireMagic™ Magbot Ablation Catheter for rapid arrhythmia (Experimental): Multicentre, target value method, single-arm
  Interventions: Device: FireMagic™ Magbot Ablation Catheter

INTERVENTIONS:
Device: FireMagic™ Magbot Ablation Catheter — All patients signed informed consent forms, enrolled in the trial, underwent surgical treatment for rapid arrhythmia using XX, and were discharged after follow-up data collection. The total duration for each subject is estimated to be approximately 7 days.

SUMMARY:
Clinical study on the safety and efficacy of FireMagic™ Magbot Ablation Catheter for rapid arrhythmia

DETAILED DESCRIPTION:
Explore the safety and efficacy of ireMagic™ Magbot Ablation Catheter for rapid arrhythmia in clinical studies, establish standards for standardised catheter use after market launch, and provide evaluation indicators that meet the requirements for nationwide multi-centre promotion.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients aged 18 to 80 years old, with no gender restrictions; 2) Patients clinically diagnosed with paroxysmal atrial fibrillation or symptomatic supraventricular tachycardia: i. For patients with paroxysmal atrial fibrillation, atrial fibrillation was recorded by surface electrocardiogram or Holter monitoring (including single-lead electrocardiogram) within one year prior to enrolment; ii. For patients with symptomatic supraventricular tachycardia, PSVT (AVNRT or AVRT) was recorded by electrocardiogram, Holter monitoring, or electrophysiological examination; 3) Patients who have not responded adequately to or are intolerant of at least one antiarrhythmic drug, or who are willing to undergo ablation surgery without prior medication; 4) Patients who fully understand the treatment plan, voluntarily sign the informed consent form, and are willing to undergo the examinations, surgery, and follow-up required by the plan.

Exclusion Criteria:

* 1) Left atrial thrombus (not applicable for PSVT); 2) Left atrial anteroposterior diameter ≥55 mm (not applicable for PSVT); 3) Left ventricular ejection fraction (LVEF) ≤40%; 4) Previous history of atrial septal defect repair or atrial myxoma (not applicable for PSVT); 5) Presence of active implantable devices (e.g., pacemaker, ICD, etc.); 6) NYHA functional class III-IV; 7) History of cerebrovascular disease within the past 6 months (including cerebral haemorrhage, stroke, transient ischaemic attack); 8) History of cardiovascular events within the past 3 months (including acute myocardial infarction, coronary artery intervention or bypass surgery, artificial valve replacement or repair, atrial or ventricular incision); 9) Acute or severe systemic infection; 10) Patients with severe liver or kidney disease, malignant tumours, or end-stage diseases, or those whom the investigator believes may interfere with the treatment, evaluation, or compliance of this trial; 11) Patients with a significant tendency to bleed, hypercoagulable states, or severe haematological disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate success rate of surgery | On the day of the surgery
  1. For patients with supraventricular tachycardia:
     Following the procedure, the following criteria are used to evaluate whether catheter ablation has achieved the intended surgical objectives:Ⅰ. AVNRT: AVNRT cannot be induced after ablation. If skipped beats or 1-2 atrial echoes are present, induction stimulation must be performed concurrently with an isoproterenol challenge test, and AVNRT still cannot be induced. Ⅱ.AVRT: ① AVRT cannot be induced after ablation; ② ventricular stimulation shows central VA Wenckebach conduction or VA dissociation; ③ atrial stimulation shows central AV Wenckebach conduction.
  2. For patients with paroxysmal atrial fibrillation:
  Observe for 20-30 minutes after initial pulmonary vein isolation and verify successful bidirectional block.

OTHER OUTCOMES:
Safety metrics: Calculate the incidence rate of adverse events associated with the use of the study device during the perioperative period. | Statistics Perioperative
  Calculate the incidence rate of any major adverse events occurring within 7 days after each atrial fibrillation ablation procedure (including initial and repeat procedures) using the study device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China